CLINICAL TRIAL: NCT06772870
Title: A Phase 1, Double-Masked, Randomized, Placebo-Controlled, Single Ascending Dose Crossover Study to Assess the Safety, Tolerability, and Pharmacokinetics of Subcutaneous and Intravenous DT-216P2 in Normal Healthy Participants
Brief Title: A Single Ascending Dose Study of DT-216P2 in Normal Healthy Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Design Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DTX-216P2-011
Record Dates: First submitted 2025-01-06; First posted 2025-01-14 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DT-216P2 (Experimental)
  Interventions: Drug: DT-216P2
- Placebo (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: DT-216P2 — DT-216P2 will be administered as subcutaneous injection, subcutaneous infusion and intravenous infusion.
  Arms: DT-216P2
Drug: Saline — Normal saline solution will be used as placebo control.
  Arms: Placebo

SUMMARY:
This purpose of the study is to evaluate the safety, tolerability and pharmacokinetics of single ascending doses of DT-216P2 administered either subcutaneously (SC) and intravenously (IV) in normal healthy participants. Approximately 36 participants will be enrolled into this study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18-45 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and ECG.
* Agree to abstain from strenuous physical activity outside of daily norm, until end of study.
* Body mass index between 16 and 32 kg/m2 (inclusive) at screening; weight should be <= 100 kg at screening.
* Male and/or female using protocol defined and regulatory approved contraception.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Any concomitant medical condition that in the opinion of the investigator, puts the participant at risk or precludes participant from completing the study protocol.
* Any clinically significant nonmedical conditions and psychiatric disorders that could put the participant at higher risk for participation in the study, influence the participant's ability to participate in the study, or interfere with interpretation of the participant's study results, in the opinion of the investigator.
* Is not willing to comply with the contraceptive requirements during the study period, as per protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of treatment emergent adverse events (TEAEs) | From first dose to end of study, Day 30 post first dose administration.
  To evaluate the safety and tolerability of single ascending doses of DT-216P2 in normal healthy participants by frequency of treatment-emergent adverse events (TEAEs).

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of DT-216P2 | Pre-dose and up to 240 hours post first dose for both SC and IV infusion.
Time to Maximum Plasma Concentration (Tmax) of DT-216P2 | Pre-dose and up to 240 hours post first dose for both SC and IV infusion.
Area Under the Concentration-time Curve (AUC) of DT-216P2 | Pre-dose and up to 240 hours post first dose for both SC and IV infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Gronen, MD, Principal Investigator — Nucleus Network
Locations (1):
- Nucleus Network, Level 5, 89 Commercial Road, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No